CLINICAL TRIAL: NCT01014559
Title: Study of Efficacy of OXN PR, Compared to Oxy PR, for Reduction of Intensity of Opioid-induced Constipation Symptoms in Pts Treated for Cancer or Non-cancer Pain: A Randomised, Double-blind, Controlled, Multicentre Study
Brief Title: Efficacy of Oxycodone/Naloxone(OXN), Versus Oxycodone (OXY), for the Reduction of Intensity of Opioid-induced Constipation in Pain Patients
Acronym: OXN3505
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Mundipharma SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXN3505; 2009-012051-20
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Constipation; Pain
Keywords: Constipation; Oxycodone; Oxycodone hydrochloride; Naloxone hydrochloride; Naloxone
MeSH Terms: conditions — Constipation; Pain | interventions — oxycodone naloxone combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged release tablet (Active Comparator): OxyCodone Naloxone controlled release tablet
  Interventions: Drug: Oxycodone Naloxone
- Tablet (Active Comparator): Oxycodone PR Tablets
  Interventions: Drug: Oxycodone PR Tablets

INTERVENTIONS:
Drug: Oxycodone Naloxone — Oxycodone Naloxone PR Tablet taken twice daily
  Arms: Prolonged release tablet
Drug: Oxycodone PR Tablets — Oxycodone PR Tablets taken twice daily
  Arms: Tablet

SUMMARY:
The primary objective of this trial is to study the efficacy of oxycodone/naloxone prolonged release tablets (OXN PR), compared to oxycodone prolonged release tablets (Oxy PR), for the reduction of the intensity of opioid-induced constipation symptoms in patients treated for cancer or non-cancer pain.

DETAILED DESCRIPTION:
Eligible patients with documented cancer or non-cancer pain, either currently receiving a WHO step II opioid and requiring the initiation of a WHO step III opioid or currently receiving a WHO step III opioid, and having opioid-related constipation defined by either a KESS score ≥9 or the current use of laxatives (≥3 times per week), will be randomly assigned to receive either OXN PR or Oxy PR. Randomisation will be stratified on the cause of pain: cancer or non-cancer.

Any patient having completed the study and wishing to receive OXN PR afterwards may enter an optional open extension phase. During this phase, all patients will receive OXN PR and be managed as per the usual practice in the center until commercial OXN PR is available in France (with a limit of 1 year after Day 28). Adverse events will be assessed at each visit.

ELIGIBILITY:
Inclusion criteria

1. Male or female patient aged 18 years or older.
2. With cancer pain or non-cancer pain such as chronic low back pain, osteoarthritis or other.
3. Either currently receiving a WHO step II opioid and requiring the initiation of a WHO step III opioid (due to a lack of efficacy of the step II opioid) expected to last 28 days or more, or currently receiving a WHO step III opioid expected to last further 28 days or more.
4. Having opioid-related constipation defined by either a KESS score ≥ 9 or the current use of laxatives (at least 3 times per week).
5. Able, in the opinion of the Investigator, to comply with the study protocol.
6. Women of childbearing potential must have a negative urine pregnancy test result at inclusion (test under supervision of the investigator) and use an effective birth control method. Women of non-childbearing potential must be postmenopausal or surgically sterile (hysterectomy and/or bilateral oophorectomy).
7. Having received oral and written information about the study protocol and signed a written, informed consent to participate.

Exclusion criteria

1. Pregnancy or breastfeeding.
2. Known contraindication or hypersensitivity to oxycodone, naloxone, bisacodyl, any chemically close substance, and ingredients.
3. Clinically significant impairment of cardiovascular, respiratory, liver or kidney function disease, as determined by medical history, clinical laboratory tests, ECG results, and physical examination, that in the opinion of the Investigator may present a risk upon exposure to the study medication.
4. Known or suspected unstable brain or spinal cord metastases that may require changes in steroid treatment throughout the duration of the study.
5. Increased intracranial pressure.
6. Evidence of clinically significant gastrointestinal disease (e.g., paralytic ileus, peritoneal carcinosis), significant structural abnormalities of the gastrointestinal tract (e.g., scarring, obstruction etc) either related or not related to the underlying cancer or disease progression.
7. Rheumatoid arthritis, as co-medication may have an impact on the study results, especially if co-medication is not stable within the study.
8. Surgery completed prior to the start of the study, or planned surgery during the study that would influence pain or bowel function during the study or preclude completion of the study.
9. Cyclic chemotherapy in the two weeks before inclusion or planned during the study that has shown in the past to influence bowel function. Patients having their first cycle of chemotherapy during the 2 weeks before the inclusion visit or during the study they should not be included in the study.
10. Radiotherapy that, in the investigators opinion, would influence bowel function or pain during the study.
11. Treatment with an opioid receptor antagonist in the month preceding inclusion.
12. History of alcohol, opioid or other drug abuse.
13. Current treatment with another psychoactive drug that, in the opinion of the Investigator, may present a risk when associated with an opioid.
14. Any somatic or psychic condition that, in the opinion of the Investigator, may compromise the ability of the patient to understand and comply with the study protocol or to provide informed consent to participate.
15. Patient who participated in a clinical research involving a new chemical entity or an experimental drug within 30 days of study entry. Concurrent enrolment in another clinical trial is not permitted unless the sole purpose of the other trial at the time of the OXN3505 inclusion visit is for long-term follow-up/survival data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change of intensity of constipation symptoms, as assessed by the BFI from baseline to Day 28. The BFI is the mean value of 3 single items: Ease of defecation; Feeling of incomplete bowel evacuation; Personal judgement of constipation. | 28 days

SECONDARY OUTCOMES:
Change of BFI from baseline (bl) to Days 7,14,21. Change of PAC-SYM score from bl to Days 7,14,21,28. Change of KESS score from bl to Days 7,14,21,28. Frequency of laxative medication use between Day 0 & Day 28. Change of pain as assessed by BPI-SF | Days 7, 14 and 21

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France